CLINICAL TRIAL: NCT03363880
Title: Establishment of Regional Severe Trauma Treatment System in 100 Counties: a National Multi-center, Cluster-randomized Controlled Trial
Brief Title: Establishment of Regional Severe Trauma Management System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, baoguojiang, Dean of Peking University People's Hospital, Director of department of orthopaedic surgery of Peking University, Chairman of China trauma rescue&treatment association, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Safe China 100 county project
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Trauma; Multiple Trauma; Emergencies
Keywords: Severe trauma; Multiple trauma; Regional Trauma management system; Trauma management team
MeSH Terms: conditions — Wounds and Injuries; Multiple Trauma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The trauma treatment team will be established in the experimental group
  Interventions: Other: trauma treatment team
- control group (Active Comparator): The trauma treatment team will not be established in this group，just establish the basic experimental settings
  Interventions: Other: Basic experimental settings

INTERVENTIONS:
Other: trauma treatment team — Establishing the trauma management system included a trauma treatment team. The severe trauma treatment team will be composed by the physicians from departments of emergency, orthopedic trauma, urology, cardiothoracic surgery, neurosurgery, general surgery, anesthesiology, and ICU.
  Arms: experimental group
Other: Basic experimental settings — Establishing the trauma management system without a trauma treatment team.
  Arms: control group

SUMMARY:
To evaluate the effects of trauma treatment team establishment on the treatment of patients with severe trauma.

DETAILED DESCRIPTION:
This is a national multi-center, cluster-randomized controlled trial. This cluster-randomized controlled trial will be performed, with counties as the randomization units. The included counties will be randomized into an experimental group and a control group. A trauma treatment team will be only established in the experimental group. The in-hospital mortality rate will be compared between the experimental and control groups to investigate the effects of trauma treatment team establishment on the treatment of patients with severe trauma.

ELIGIBILITY:
In this study, three-level subjects (counties, hospitals, and trauma patients) will be included according to the following inclusion and exclusion criteria:

* inclusion:
* Inclusion criteria of counties:

  * National counties and county-level administrative regions;
  * Local government and health management department have the desire and requirements to establish a standardized trauma emergency treatment system;
  * More than 500,000 people;
  * With pre-hospital emergency treatment system;
  * Trauma first aid needs: No less than 20 patients with severe trauma (ISS ≥ 16) throughout the county;
* Inclusion criteria of hospitals:

  * With the most advanced regional treatment resources during the entire period from trauma recovery to rehabilitation for third-grade class A hospitals;
  * With basic trauma treatment resources for second-grade class A hospitals;
  * Trauma doctors are on call 24 hours a day and can participate in the early treatment of patients with trauma;
* Inclusion criteria of patients:

  * Patients with acute trauma occurring within 48 hours;
  * Patients are transferred to trauma treatment center hospital or trauma treatment non-center hospitals;
  * Patients themselves go to or are transferred by their family members to the trauma treatment center hospital or trauma treatment non-center hospita;
* Exclusion:
* Exclusion criteria of counties:

  ○ All second-grade class A or third-grade class A hospitals in the county cannot establish a trauma treatment team because of various reasons;
* Exclusion criteria of hospitals:

  ○ Hospitals can not establish a trauma treatment team because of various reasons;
* Exclusion criteria of patients:

  * Patients with trauma from regions not included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7250 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality rate | from hospital admission to discharge, an average of 20 days
  the percentage of patients who die after hospitalization for severe trauma in admitted patients with severe trauma.

SECONDARY OUTCOMES:
Mortality rate of patients with severe trauma within 30 days after trauma attack | within 30 days after trauma attack
  the percentage of patients who die within 30 days after trauma attack in admitted patients with severe trauma
Mortality rate of patients with severe trauma within 30 days after discharge | within 30 days after discharge
  the percentage of patients who die within 30 days after discharge in admitted patients with severe trauma

CONTACTS AND LOCATIONS:
Overall Officials: baoguo Jiang, MD, Principal Investigator — Peking University People's Hospital; Peking University Traffic Medical Center; China Trauma Rescue&Treatment Association

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Liu HX, Wang YH, Zhang YJ, Zhang JJ, Huang W, Jiang BG, Wang TB. Establishment of trauma treatment teams within a regional severe trauma treatment system in China: study protocol for a national cluster-randomised trial. BMJ Open. 2018 Dec 4;8(12):e023347. doi: 10.1136/bmjopen-2018-023347. PMID 30518584